CLINICAL TRIAL: NCT00766168
Title: Prospective Study of Substantial Equivalence of Rigid Gas Permeable HDS HI 1.54™ Daily Wear Lenses for Correction of Naturally Occurring Myopia and Hyperopia From +20 to - 20 D Sphere (Spectacle Plane) With and Without Astigmatism.
Brief Title: High Refractive Index Material 510(k)
Acronym: PVS-07-07
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision International Limited (CVIL) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HDSHI154; PVS-07-07
Record Dates: First submitted 2008-10-01; First posted 2008-10-03 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Myopia; Hyperopia
Keywords: contact lens; rigid gas permeable; refractive index
MeSH Terms: conditions — Myopia; Hyperopia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): FluoroPerm 30 RGP lens daily wear
  Interventions: Device: FluoroPerm 30 RGP; paflufocon C
- HDS HI 1.54 (Experimental): New rigid gas permeable contact lens material material
  Interventions: Other: HDS HI 1.54; pahrifocon A

INTERVENTIONS:
Other: HDS HI 1.54; pahrifocon A — Contact Lens
  Other Names: pahrifocon A
  Arms: HDS HI 1.54
Device: FluoroPerm 30 RGP; paflufocon C — Contact lens daily wear
  Other Names: paflufocon C
  Arms: Control

SUMMARY:
The purpose of this study is to establish the substantial equivalence of the HDS HI 1.54™ to the paflufocon C material control lenses to correct myopia and hyperopia with and without astigmatism. The purpose of the study is to profile the outcome endpoints and the patient acceptance of this Class II medical device.

DETAILED DESCRIPTION:
Seventy six (76) subjects (152 eyes) were enrolled and dispensed in the multisite, randomized, double masked clinical study to provide data that support the presumption of equivalence of the HDS HI 1.54™ investigational lenses to a historical control contact lens. Sixty four (64) subjects (84.2%) completed the study and 12 subjects (15.8%) were discontinued. The population demographics were similar to previous contact lens studies.

Of the ten Test subjects who discontinued, Difficulty Cleaning Lenses (3 subjects) and Poor Comfort (2 subjects), Poor Vision (1 subject) and Poor Vision and Poor Comfort (2 subjects) accounted for 80% of the discontinuations. Two Control subjects discontinued, one for Loss of Interest and one for Poor Comfort There were no adverse events reported during the study. The only study related complications were slit lamp findings of grade 3 for injection. Each of these resolved without complication.

Slit lamp findings were reported at frequencies within expected values and the positive slit lamp observations were primarily grade 1 (trace). Staining and injection were reported most frequently. Subject reports of no symptoms were lowest at the 1 week visit for both the Completed Test and Control eyes and then increased over the remainder of the study. Discomfort was reported most frequently (13.7% of Completed Test eye visits and 12.3% of Completed Control Eye visits). .

Lens comfort was rated as an average of 4.04 (very good) for the Completed Test eyes and 4.07 (very good) for the Completed Control eyes. This compared to a baseline value of 3.96 for the Test eyes and 4.23 for the Control eyes with the pre-study habitual correction.

Keratometry changes were within 1.00 diopter for 93.1% of the Completed Test eyes and 96.4% of the Completed Control eyes. Manifest refraction changes were within 1.00 diopter for 97.9% of the Completed Test eyes and 98.2% of the Completed Control eyes.

One eye of the 63 Completed Test eyes targeted for full distance vision was reported to show a decrease in contact lens visual acuity from the baseline best corrected visual acuity of greater than 0.20 logMAR. The reason for the loss was a reported baseline measurement error. One eye of the 48 Completed Control eyes targeted for full distance vision was reported to show a decrease in contact lens visual acuity from the baseline best corrected visual acuity of greater than 0.20 logMAR. The reason cited for the decrease was lenses being switched eye for eye.

Average lens wearing time was stable at over 13 hours per day for the Completed Test and Control subjects and showed a decrease over time for the discontinued eyes.

Forty nine (49) lens replacements were made for 40 of the 152 eyes dispensed in the study. The replacements were predominantly for deposits (8) or parameter and power change (21) which together account for 59% of the lens replacements. Discomfort was cited for 18.4% (5 test and 4 control lenses) of the lens replacements. Five lenses (10%) were replaced due to loss.

The results of the clinical evaluation of the Paragon HDS HI 1.54™ contact lenses provide evidence of substantial equivalence to the historical control, Paragon Fluroperm® 30 contact lenses.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects may be male or female, of any race, and at least 12 years old at the time of the pre-treatment examination.
2. The prospective eye(s) must have naturally occurring refractive myopia up to -20.00 D or hyperopia or aphakia up to +20.00 D sphere (spectacle plane), with less than 10.00 D of refractive astigmatism (spectacle plane), as determined by manifest refraction (phoropter or trial frame with a 12.5 mm vertex distance). Subjects must have best spectacle corrected visual acuity of at least 0.30 logMAR (20/40) in each eye.
3. All subjects must be treated bilaterally.
4. Subjects must be willing and capable to return for all scheduled follow-up visits for a period of at least 3 months.

Exclusion Criteria:

1. Female subjects who are pregnant, breast-feeding or intend to become pregnant over the course of the study.
2. Subjects with a history of any of the following medical conditions: collagen vascular disease, autoimmune disease, immunodeficiency diseases, ocular herpes zoster or simplex, endocrine disorders (including, but not limited to active thyroid disorders and diabetes), lupus, and rheumatoid arthritis.

   NOTE: The presence of diabetes (either type 1 or 2), regardless of disease duration, severity or control, will specifically exclude subjects from eligibility.
3. Subjects with a history of intraocular or corneal surgery (excluding cataract extraction and refractive surgery), active ophthalmic disease or abnormality (including, but not limited to, blepharitis, recurrent corneal erosion, dry eye syndrome, neovascularization > 1mm from limbus), clinically significant lens opacity, clinical evidence of trauma (including scarring), or with evidence of glaucoma or propensity for narrow angle glaucoma as determined by gonioscopic examination in either eye.

   NOTE: This includes any patient with open angle glaucoma, regardless of medication regimen or control. Additionally, any patient with an IOP greater than 21 mm Hg at baseline is specifically excluded from eligibility.
4. Subjects with evidence of keratoconus, corneal irregularity, or abnormal videokeratography in either eye.
5. Subjects who are participating in any other clinical trial (FDA or other).

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2008-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity vs Control | 3 months
  Of the 72 Completed Test eyes, seven (7) eyes were reported to show a decrease in visual acuity of greater than 0.20 logMAR of which six (6) eyes were for a targeted monovision near power. Of the 56 Completed Control eyes eight (8) eyes were reported to show a decrease in visual acuity of greater than 0.20 logMAR of which seven (7) eyes were for a targeted monovision near power. The reasons cited for the decrease of the remaining Test eye was a reported baseline measurement error and for the remaining Control eye was lenses being switched eye for eye.

SECONDARY OUTCOMES:
Incidence of problems , symptoms and complaints vs control | 3 months
  For the Completed Test eyes, no symptoms were reported for 23.0% (107/466) of the eye symptom reports after the baseline visit. For the Completed Control eyes, no symptoms were reported for 28.6% (100/350) of the eye symptom reports after the baseline visit. For Discontinued Test eyes no symptoms were reported at 13.2% (10/76) of the eye symptom reports while the Discontinued Control eyes reported no symptoms at 15% (3/20) of the eye symptom reports.
slit lamp observations greater than grade 3 | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jerome A. Legerton, OD, MS, Study Director — Consultant to Paragon Vision Sciences
Locations (8):
- United States (8):
  - Mission Optometry, Lake Elsinore, California
  - Eyecare Consultants, Englewood, Colorado
  - Vision Care Associates, East Lansing, Michigan
  - Koetting Associates, St Louis, Missouri
  - Visionary Eye Associates, Rochester, New York
  - Western Reserve Vision Care, Beachwood, Ohio
  - Choate Eye Associates, Goodlettsville, Tennessee
  - Twin Lakes Vision Clinic, Federal Way, Washington